CLINICAL TRIAL: NCT05947916
Title: Effect of Real Time Continuous Glucose Monitoring System on Management of Women With Type 2 Diabetes Mellitus During Pregnancy in a Multidisciplinary Comprehensive System
Brief Title: Real Time Continuous Glucose Monitoring System in T2DM With Pregnacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2DMCGMs
Record Dates: First submitted 2023-03-26; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-03

CONDITIONS: Type2diabetes; Pregnancy Related; Continuous Glucose Monitoring; Time in Range; Pregnancy Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will wear real-time CGM (120 cases) to monitor blood glucose and is required to use real-time-CGM more than 50% of the time every 4 weeks, the more the better.
  Interventions: Device: Real-time Continuous Glucose Monitoring System
- Control group (No Intervention): The control group will be followed up with traditional SMBG (120 cases) monitoring.

INTERVENTIONS:
Device: Real-time Continuous Glucose Monitoring System — The intervention group wore real-time CGM (120 cases) to monitor blood glucose, and was required to use real-time-CGM more than 50% of the time every 4 weeks, the more the better.
  Arms: Intervention group

SUMMARY:
The prevalence of type 2 diabetes mellitus (T2DM) in women of childbearing age is increasing rapidly, and low glucose compliance leads to an increased risk of adverse pregnancy outcomes for mothers and infants during pregnancy in women with T2DM. Real-time continuous glucose monitoring (CGM) is an important tool for glucose monitoring and patient education, as it can continuously record blood glucose throughout the day and provide real-time feedback on high and low blood glucose levels. This is a multicenter, open-label, randomized controlled clinical study to investigate the efficacy, safety, and maternal and infant pregnancy outcomes of using real-time CGM monitoring compared with conventional self-monitoring of blood glucose (SMBG) on the basis of multidisciplinary management in pregnant women with T2DM. One hundred and twenty pregnant women with T2DM in early pregnancy who were enrolled in intensive insulin therapy were randomly divided into the real-time CGM group and the conventional SMBG group. The real-time CGM intervention group wore real-time CGM for more than 50% of the pregnancy in addition to regular SMBG; the control group only performed regular SMBG. Both groups wore Medtronic iPro 2 for 3 days in early, mid and late pregnancy, and the time in the target range of blood glucose (TIR) was recorded in a blinded manner. Primary outcome: differences in TIR between the two groups of pregnant women in early, mid, and late pregnancy. Secondary outcomes included differences in glycated hemoglobin, hypoglycemia, insulin dose before delivery, pregnancy weight gain, and maternal and infant pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A clear history of type 2 diabetes, or a history of type 2 diabetes diagnosed in early pregnancy
* Singleton gestation at 4-12 weeks, with substandard glycemic control (i.e., fasting glucose > 5.3 mmol/L, and or 1 hour postprandial glucose > 7.8 mmol/L, and or 2 hours postprandial glucose > 6.7 mmol/L) after lifestyle intervention ± basal insulin therapy, as assessed by the endocrinology department. Patients who need insulin regimen with basal plus meal or insulin pump regimen.
* Patients are willing and committed to establish and follow up in the obstetrics and gynecology departments of Peking University Third Hospital, Haidian District Hospital and Yanqing District Hospital during pregnancy, and are willing to provide information on obstetric examination and perinatal medical records if they are transferred to the hospital for special reasons for follow-up or delivery.
* Voluntarily participate in the study, examine and follow up according to this project and sign informed consent.
* Able to pass the screening period Adherence evaluation

Exclusion Criteria:

* Patients with type 1 diabetes, specific type of diabetes or gestational diabetes
* Pregnancy with severe comorbidities or diabetic complications for which obstetrics does not recommend continuation of pregnancy, including but not limited to the following: proliferative retinopathy, chronic kidney disease (eGFR less than 60 mL/min/1.73± massive proteinuria), known coronary and cerebrovascular disease, autoimmune system disease and receiving exogenous glucocorticoids or immunosuppressive therapy.
* Patients who have been hospitalized for psychiatric treatment within 6 months prior to enrollment or are still on psychiatric medications.
* Patients who have received other interventional studies.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of Time in Range (TIR) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The iPro2 device was used to calculate TIR(the control range of blood glucose during pregnancy was 3.5-7.8mmol/L), and the average value of TIR obtained from two measurements was used as the main outcome index.

SECONDARY OUTCOMES:
Time Above Range(TAR） | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2(the time above control range of blood glucose during pregnancy)
Time Below Range(TBR) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2 (the time below control range of blood glucose during pregnancy)
Mean Amplitude Of Glycemic Excursion(MAGE) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Coefficient of Variation (CV) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Standard difference (SD) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Mean absolute relative difference (MARD) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Interquartile range(IQR) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Interdencile range (IDR) | 24-28 weeks (second trimester), 34-38 weeks (2 weeks before delivery)
  The data were recorded via iPro2.
Patient-reported severe hypoglycemic events | From enrollment to 42 weeks gestation
  Number of patient-reported severe hypoglycemic events (hypoglycemic events requiring assistance) from enrollment to 42 weeks of gestation.
Patient-reported severe hypoglycemic events | From enrollment to 42 weeks gestation
  (a) Number of patient-reported severe hypoglycemic events (hypoglycemic events requiring assistance) from enrollment to 42 weeks of gestation; (b) Number of mild hypoglycemic (<3.5 mmol/l) and moderate hypoglycemic (<2.8 mmol/L) events detected by patient self-monitoring from enrollment to 42 weeks of gestation (c) Area under the curve for mild hypoglycemia (<3.5 mmol/l) and moderate hypoglycemia (<2.8 mmol/L) at 24, 28 and 34 weeks of gestation as indicated by the ambulatory glucose monitoring device; (d) Area under the curve for mild hypoglycemia (<3.5 mmol/l) and moderate hypoglycemia (<2.8 mmol/L) at night (23:00-7:00) as indicated by the ambulatory glucose monitoring device at 24, 28 and 34 weeks of gestation.
Number of moderate hypoglycemic events | From enrollment to 42 weeks gestation
  Number of moderate hypoglycemic (<2.8 mmol/L) events detected by patient self-monitoring from enrollment to 42 weeks of gestation; Area under the curve for moderate hypoglycemia (<2.8 mmol/L) at 24, 28 and 34 weeks of gestation as indicated by the ambulatory glucose monitoring device; (d) Area under the curve for moderate hypoglycemia (<2.8 mmol/L) at night (23:00-7:00) as indicated by the ambulatory glucose monitoring device at 24, 28 and 34 weeks of gestation.
Number of mild hypoglycemic events | From enrollment to 42 weeks gestation
  Number of mild hypoglycemic (<3.5 mmol/l) events detected by patient self-monitoring from enrollment to 42 weeks of gestation (c) Area under the curve for mild hypoglycemia (<3.5 mmol/l) at 24, 28 and 34 weeks of gestation as indicated by the ambulatory glucose monitoring device; (d) Area under the curve for mild hypoglycemia (<3.5 mmol/l) at night (23:00-7:00) as indicated by the ambulatory glucose monitoring device at 24, 28 and 34 weeks of gestation.
Total insulin | At 4 weeks after enrollment, 24, 28, 34 weeks gestation and 6 weeks postpartum.
  the whole day dose of insulin
Maternal weight gain | From enrollment to 42 weeks gestation
  The absolute value of maternal weight gain during pregnancy
Glycosylated hemoglobin | During delivery
  Glycosylated hemoglobin during delivery
Glycosylated albumin | During delivery
  Glycosylated albumin during delivery
Number of Patients with Adverse pregancy outcome | 6 weeks postpartum.
  Includign gestational hypertension, preeclampsia/eclampsia, Cesarean section rate, puerperal infection.
Number of Pregnancy loss | From enrollment to 6 weeks postpartum.
  Including abortion (less than 28 weeks gestation), stillbirth and neonatal death.
Apgar score | During delivery
  Apgar score at birth, range from 0-10, evaluated activity, pulse, grimace, appearance, respiration. Score 8 to 10 is classified as no asphyxia, 4 to 7 is mild asphyxia, 0 to 3 is severe asphyxia
Number of neonatal hypoglycemia | 6 weeks postpartum.
  Intravenous glucose infusion is required.
The length of a newborn is treated in the neonatal intensive care unit (NICU) | 6 weeks postpartum.
  The length of a newborn is treated in the neonatal intensive care unit (NICU)
Gestational age at birth | During delivery
  The incidence of preterm delivery (28-37 weeks gestation at birth), full-term delivery (37-42 weeks gestation at birth), and overdue delivery (more than 42 weeks gestation at birth).
Number of macrosomia or fetal growth restriction | During delivery
  Macrosomia (birth weight greater than 4000 g) or fetal growth restriction (birth weight less than 2500)
Number of newborns with neonatal birth injury, shoulder dystocia, neonatal jaundice, neonatal respiratory distress syndrome (RDS) | From birth to discharge.
  Including neonatal birth injury, shoulder dystocia, neonatal jaundice, neonatal respiratory distress syndrome (RDS).

OTHER OUTCOMES:
Security Index | From enrollment to 6 weeks postpartum.
  Outpatient and emergency treatment of patients for any reason (except planned follow-up), record the number of visits, cause, diagnosis and corresponding treatment.
Security Index-Medication other than insulin during pregnancy. | From enrollment to 6 weeks postpartum.
  Medication other than insulin during pregnancy.
Adverse event record | From enrollment to 6 weeks postpartum.
  Adverse events other than those described above.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No